CLINICAL TRIAL: NCT04813094
Title: An Internet-Based Integrated-management Program to Control Readmission and Health-related Quality of Life Among Patients With Atrial Fibrillation: a Randomized Controlled Trial
Brief Title: An Integrated-management Program to Control Health-related Quality of Life Among Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Fung-Wei Chang, Director, Head of Obstetrics and Gynecology, Clinical Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tri_20210311
Record Dates: First submitted 2021-03-11; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation
Keywords: Internet-Based; Atrial fibrillation; readmission; health-related quality of life
MeSH Terms: conditions — Atrial Fibrillation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Based integrated-management Program (Experimental): The Internet-based integrated management Program system have five domains that included patient's information collection, AF knowledge area, instructions on anticoagulation medicine, self-monitoring of symptom area, and professional consultation. Participants will have their own account and passwords to log in to the system via mobile phones or computers. Everyone will have their own area to ensure the privacy of participants. The research nurse will have sent messages every day to care about the participant's condition.
  Interventions: Other: Internet-Based integrated-management Program
- Control group (Active Comparator): Patients in the control group will receive standard nurse consultations and three-time telephone coaching.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Internet-Based integrated-management Program — The Internet-based integrated management Program system have five domains that included patient's information collection, AF knowledge area, instructions on anticoagulation medicine, self-monitoring of symptom area, and professional consultation. Everyone have their own area to ensure the privacy of participants. The research nurse has sent messages every day to care about the participant's condition. In this area, when the participant have an emergency, it not only provided textual information, but also provided telephone coaching.
  Arms: Internet-Based integrated-management Program
Other: Control group — Patients in the control group will receive standard nurse consultations and three-time telephone coaching.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effectiveness of the Internet-based integrated-management Program on increasing coping strategies, medical adherence and HRQoL, and reducing readmission in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Design a double-blind two-group longitudinal experimental study will be conducted to compare the Internet-based integrated-management Program with a usual care.

After receiving informed consents, participants will be randomly assigned to two groups by using a web-based system with blocked randomization. The intervention group will receive an Internet-based integrated management Program, and control group will receive nurse consultations and three times telephone coaching. Outcomes from three self-report questionnaires at 1 month, 3 months and 6 months after initiating the intervention will be compared to baseline assessments. Outcome measurements include the following parameters: 28-item Brief COPE, Medication Adherence Rating Scale (MARS), the 3-level version of EuroQol five-dimension self-report questionnaire (EQ-5D-3L), and readmission events.

Inclusion and exclusion criteria: The inclusion criteria are: (1) those who are ≥20 years old and AF diagnosed by a cardiology specialist, (2) have clear consciousness, (3) are fluent in Mandarin/Taiwanese, (4) are receiving anticoagulant treatment, (5) are able to use mobile phone and compute. The exclusion criteria are: (1) diagnosed with any psychiatric disorder, (2) are involved in other clinical trials.

Recruitment Participants will be recruited from a cardiology outpatient clinic of a medical center in northern Taiwan. The study design and protocols had been reviewed and approved by the institutional review board of the participating hospital. At the content session, all assessments and procedures will be fully explained.

Assessment of eligibility and randomization: Participants will be considered eligible if they meet the inclusion criteria. All participants will be informed that they are able to withdraw from the study at any time. Before randomization, participants will be asked to answer four questionnaires. The questionnaires include demographic characteristics, 28-item Brief COPE, Cardiac Symptom Survey (CSS), Medication Adherence Rating Scale (MARS), and the 3-level version of EuroQol five-dimension self-report questionnaire (EQ-5D-3L).

Double blinding is maintained because i) research nurse who is involved in the collection of post-test data are not having any information of group assignment. ii) Participants do not know their group assignment and receive corresponding interventions.

The Internet-based integrated management Program is conducted in the cardiology outpatient department. Participants will have their own account and passwords to log in to the system via mobile phones or computers. The system has five domains that included patient's information collection, AF knowledge area, instructions on anticoagulation medicine, self-monitoring of symptom area, and professional consultation. Everyone has their own area to ensure the privacy of participants. The research nurse will have sent messages every day to care about the participant's condition. In this area, when the participants have an emergency, it will not only provide textual information, but also provide telephone coaching. In addition, the investigators also will instruct participants and provide the AF management manual, which will include a description of the causes and predisposing risk factors of AF, the symptoms of AF, the relationship between AF and stroke, stroke prevention measures for patients with AF, and managing a healthy lifestyle.

Patients in the control group will receive standard nurse consultations. A manual of AF management is provided and explained. In addition, the investigators will provide a three-time telephone coaching, which will teach participants how to manage their disease and associated disease knowledge at the 1 month, 3 months and 6 months after random assignment.

Coping strategies: The 28-item Brief COPE self-report questionnaire measure strategies participants use for coping. The Brief-COPE is divided into approach coping, in which individuals actively seek resources to deal with their health problems; and avoidance coping, in which individuals attempt to divert attention away from events. Higher scores indicate greater use of the specific coping strategy.

Medicine adherence: This 10-items MARS scale has three domains: medication adherence behavior, attitude toward taking medication, and negative side-effects and attitudes to medication. The total possible score ranged from 0 to 10. A higher score indicates a better medicine adherence.

Health-Related Quality of Life: Participant's HRQoL was measured by the 3-level version of EuroQol five-dimension self-report questionnaire (EQ-5D-3L). The instrument has two subscales: the EQ-5D descriptive system (5 items) and the EuroQol visual analog scale (EQ-VAS). The EQ-5D descriptive system have five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. EQ-VAS is an individual's self-assessment of health status, with a vertical scale of 20 cm (visual analog scale). The higher score indicates the best possible state of health.

Readmission events: After inclusion in the study, the investigators will follow up readmission events in all included participants. The readmission events are based on the query of medical records in the research hospital.

Statistical analysis: the investigators will use descriptive statistics (mean, standard deviation, frequency and percentage) to analyze participant characteristics and outcomes. The initial differences between groups for demographic characteristics, coping strategies, medical adherence, and HRQoL will be examined with independent t-tests and Chi-square analysis. Effects of the Internet-based integrated-management Program on coping strategies, medical adherence, and HRQoL in patients with AF will be analyze using generalized estimating equations (GEE). The significance will be defined as a two-tailed P-value of < 0.05.

Patient's characteristics will report as age, gender, type of AF, the class of mEHRA, comorbidities and medication status are evaluated by the univariate logistic regression to assess the association with the readmission events. Predictor variables with P value <0.20 are eligible for inclusion in the multivariable logistic regression model for the outcome. The continuous variables are converted to categorical variables in the multivariable logistic model. In the multivariable logistic regression model, predictor variables with two-tailed P value <0.05 are considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Atrial fibrillation
2. ≥20 years old
3. Have a clear consciousness
4. Fluent in Mandarin/Taiwanese
5. Receiving anticoagulant treatment
6. Able to use mobile phones and computers.

Exclusion Criteria:

1. Psychiatric disorder
2. Participate in other clinical trials.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Coping strategies | Change from coping strategies at 1 months, 3 months and 6 months.
  The 28-item Brief COPE self-report questionnaire measure strategies participants use for coping. The Brief-COPE is divided into approach coping, in which individuals actively seek resources to deal with their health problems; and avoidance coping, in which individuals attempt to divert attention away from events. Higher scores indicate greater use of the specific coping strategy.
Medicine adherence | Change from medicine adherence at 1 months, 3 months and 6 months.
  This 10-items MARS scale has three domains: medication adherence behavior, attitude toward taking medication, and negative side-effects and attitudes to medication. The total possible score ranged from 0 to 10. A higher score indicates a better medicine adherence.
Health-Related Quality of Life | Change from Health-Related Quality of Life at 1 months, 3 months and 6 months.
  Participant's HRQoL was measured by the 3-level version of EuroQol five-dimension self-report questionnaire (EQ-5D-3L). The instrument has two subscales: the EQ-5D descriptive system (5 items) and the EuroQol visual analog scale (EQ-VAS). The EQ-5D descriptive system have five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. EQ-VAS is an individual's self-assessment of health status, with a vertical scale of 20 cm (visual analog scale). The higher score indicates the best possible state of health.

SECONDARY OUTCOMES:
Readmission events | Change from readmission events at after intervention within 2 years.
  After inclusion in the study, we will follow up readmission events in all included participants. The readmission events are based on the query of medical records in the research hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Kao, PHD, Study Director — Taiwan Nurses Association
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] Pistoia F, Sacco S, Tiseo C, Degan D, Ornello R, Carolei A. The Epidemiology of Atrial Fibrillation and Stroke. Cardiol Clin. 2016 May;34(2):255-68. doi: 10.1016/j.ccl.2015.12.002. Epub 2016 Mar 18. PMID 27150174
- [Result] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Result] Tse HF, Wang YJ, Ahmed Ai-Abdullah M, Pizarro-Borromeo AB, Chiang CE, Krittayaphong R, Singh B, Vora A, Wang CX, Zubaid M, Clemens A, Lim P, Hu D. Stroke prevention in atrial fibrillation--an Asian stroke perspective. Heart Rhythm. 2013 Jul;10(7):1082-8. doi: 10.1016/j.hrthm.2013.03.017. Epub 2013 Mar 15. PMID 23501173
- [Result] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Result] Krijthe BP, Kunst A, Benjamin EJ, Lip GY, Franco OH, Hofman A, Witteman JC, Stricker BH, Heeringa J. Projections on the number of individuals with atrial fibrillation in the European Union, from 2000 to 2060. Eur Heart J. 2013 Sep;34(35):2746-51. doi: 10.1093/eurheartj/eht280. Epub 2013 Jul 30. PMID 23900699
- [Result] Chiang CE, Wang KL, Lin SJ. Asian strategy for stroke prevention in atrial fibrillation. Europace. 2015 Oct;17 Suppl 2:ii31-9. doi: 10.1093/europace/euv231. PMID 26842113
- [Result] Chiang CE, Wu TJ, Ueng KC, Chao TF, Chang KC, Wang CC, Lin YJ, Yin WH, Kuo JY, Lin WS, Tsai CT, Liu YB, Lee KT, Lin LJ, Lin LY, Wang KL, Chen YJ, Chen MC, Cheng CC, Wen MS, Chen WJ, Chen JH, Lai WT, Chiou CW, Lin JL, Yeh SJ, Chen SA. 2016 Guidelines of the Taiwan Heart Rhythm Society and the Taiwan Society of Cardiology for the management of atrial fibrillation. J Formos Med Assoc. 2016 Nov;115(11):893-952. doi: 10.1016/j.jfma.2016.10.005. Epub 2016 Nov 24. PMID 27890386
- [Result] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Derived] Hsieh HL, Kao CW, Cheng SM, Chang YC. A Web-Based Integrated Management Program for Improving Medication Adherence and Quality of Life, and Reducing Readmission in Patients With Atrial Fibrillation: Randomized Controlled Trial. J Med Internet Res. 2021 Sep 22;23(9):e30107. doi: 10.2196/30107. PMID 34550084